CLINICAL TRIAL: NCT07097519
Title: Effects on Anxiety, Stress, and Work Performance of Intensive Care Nurses Using an Immersive Virtual Reality Application
Brief Title: Effects of Virtual Reality on Anxiety, Stress, and Work Performance in ICU Nurses
Acronym: VR-ICU Nurse S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve BEKE, Phd, Nurse Educator, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-292
Record Dates: First submitted 2025-07-25; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Stress; Performance; Immersive Virtual Reality; Intensive Care (ICU); Nurse
Keywords: Job Performance; Immersive Virtual Reality; Intensive Care Nursing

STUDY DESIGN:
Intervention Model Description: This study uses a single-group, prospective, interventional, pre-test-post-test design. All participants receive the same immersive virtual reality (IVR) intervention without a comparison or control group. The intervention consists of regular use of a commercially available VR exergame (Beat Saber) for a minimum of 10 minutes per session over an 8-week period. Measurements are taken at three time points (baseline, mid-intervention, and post-intervention) using validated scales for anxiety, stress, job performance, and satisfaction. This model allows assessment of within-subject changes over time in response to the VR-based stress management and performance-enhancement intervention.
Masking Description: This study does not involve masking. It is an open-label, single-group intervention, and both participants and researchers are aware of the intervention being administered. Therefore, no additional parties are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immersive Virtual Reality Intervention for ICU Nurses (Experimental): Participants in this arm are registered nurses working in an intensive care unit who receive an immersive virtual reality (IVR) intervention. The intervention involves the use of a VR exergame (Beat Saber) through Oculus Quest 2 headsets. Nurses engage in VR sessions for a minimum of 10 minutes per day across 8-16 clinical workdays over an 8-week period. The intervention is designed to reduce anxiety and stress levels and enhance job performance. Outcome measures include anxiety, stress, individual job performance, and satisfaction ratings collected pre- and post-intervention.
  Interventions: Other: Immersive Virtual Reality (IVR)

INTERVENTIONS:
Other: Immersive Virtual Reality (IVR) — This intervention involves the use of a high-end immersive virtual reality (IVR) application through the Oculus Quest 2 headset. Nurses participate in a rhythm-based exergame, Beat Saber, for at least 10 minutes per session, during 8-16 clinical shifts over an 8-week period. The game engages users in physical movement to music, requiring whole-body coordination and providing visual, auditory, and haptic feedback. The intervention aims to reduce stress and anxiety and enhance job performance among ICU nurses by providing an immersive, engaging, and therapeutic experience within the clinical environment.

SUMMARY:
Intensive care unit (ICU) nurses often experience high levels of stress and anxiety due to the emotional demands of caring for critically ill patients. These psychological burdens can negatively affect their job performance and the quality of care they provide. Recent studies suggest that immersive virtual reality (IVR) technology may help reduce stress and improve professional performance among healthcare workers. However, no study to date has specifically evaluated the effects of IVR on ICU nurses' anxiety, stress, and job performance.

This study aims to evaluate whether an IVR application can reduce anxiety and stress levels while enhancing the job performance of ICU nurses. By introducing a clinical intervention based on virtual reality, the research seeks to explore its potential as a practical tool in improving nurses' well-being and work effectiveness in high-pressure environments. The findings will contribute to understanding the clinical applicability of IVR as a stress-reduction and performance-enhancement method in intensive care settings.

DETAILED DESCRIPTION:
This study investigates the impact of an immersive virtual reality (IVR) intervention on the anxiety, stress, and professional performance of registered nurses working in intensive care units (ICUs). ICU nurses frequently face emotionally demanding situations, including end-of-life care, which can lead to elevated stress and anxiety levels. These psychological challenges have been associated with decreased job performance and compromised quality of patient care.

Technological innovations, particularly in virtual reality, offer promising solutions for mental health support and professional development in healthcare. IVR has been used successfully in various healthcare settings to reduce stress, improve coping strategies, and enhance performance. Despite this, no study has yet specifically examined its effect on ICU nurses.

In this randomized controlled trial, participants will be assigned to either an intervention group using the IVR application or a control group receiving standard care. The IVR experience is designed to promote relaxation, reduce psychological strain, and reinforce professional competencies through immersive scenarios. Outcome measures will include validated scales for anxiety, stress, and job performance, collected before and after the intervention.

The ultimate goal of this study is to assess the clinical applicability of IVR technology in supporting ICU nurses' mental well-being and work performance, offering a novel approach to workforce resilience in critical care settings.

ELIGIBILITY:
Inclusion Criteria:

* Willing to voluntarily participate in the study
* Currently employed as a nurse in the Anesthesia and Reanimation Intensive Care Unit
* Has been working in the unit for at least 3 months
* Able and available to use the virtual reality (VR) application for a minimum of 10 minutes per day
* Willing to use the VR application on 8 to 16 clinical workdays during the 8-week intervention period

Exclusion Criteria:

* Any condition that prevents communication, completing questionnaires, or participating in measurements
* Physical limitations that prevent movement (e.g., amputation, joint restriction)
* Health problems that interfere with VR use, including chronic pain, hearing or vision loss, migraine, vertigo, nausea, epilepsy, claustrophobia, head injuries, or psychiatric treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Job Performance Measured by the Individual Work Performance Scale | From enrollment to the end of treatment at 8 weeks
  Job performance will be assessed using the Turkish version of the Individual Work Performance Scale adapted by Köroğlu Kaba & Öztürk (2021). The 14-item scale includes 3 subscales: Task Performance (5 items), Contextual Performance (6 items), and Counterproductive Work Behavior (3 items, reverse-coded). Items are rated on a 5-point Likert scale from 1 (Rarely) to 5 (Always). Higher scores indicate better performance. The internal consistency of the total scale is reported as 0.80.

SECONDARY OUTCOMES:
Change in Anxiety Level | Before and after each VR session, from enrollment to the end of treatment at 8 weeks
  Anxiety levels will be measured using the Spielberger State Anxiety Scale (STAI-State), a validated 20-item self-report questionnaire. The scale evaluates how participants feel at a specific moment, with scores ranging from 20 to 80. Higher scores indicate higher anxiety. The primary analysis will compare pre- and post-intervention scores to evaluate the effect of the immersive virtual reality (IVR) application on anxiety reduction among ICU nurses.
Change in Anxiety Levels Measured by the Spielberger State Anxiety Scale | From enrollment to the end of treatment at 8 weeks
  Anxiety levels will be assessed using the Turkish version of the Spielberger State Anxiety Scale (STAI-State), a 20-item self-report scale that measures how the participant feels in a specific moment. Each item is scored from 1 (Not at all) to 4 (Very much so), with total scores ranging from 20 to 80. Higher scores indicate greater anxiety. The scale has high internal consistency (KR-20: 0.94-0.96). It will be administered on the first and last day of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared in order to maintain participant confidentiality and comply with institutional data protection policies. The data include sensitive psychological and professional information collected from ICU nurses, which could pose privacy risks if shared.